CLINICAL TRIAL: NCT07107568
Title: Assessment of Coronary Artery Disease Before Transcatheter Aortic Valve Replacement: A Randomized, Multicenter, Non-Inferiority Trial
Acronym: TAVR-CT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1124/2025
Record Dates: First submitted 2025-07-28; First posted 2025-08-06 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Aortic Valve Stenosis and Insufficiency; Coronary Artery Disease(CAD); Transcatheter Aortic Valve Replacement (TAVR)
Keywords: TAVR-CT; PCD-CT; Severe Aortic Stenosis; Transcatheter Aortic Valve Replacement; TAVR; Photon-Counting Detector CT; Randomized Controlled Trial
MeSH Terms: conditions — Aortic Valve Stenosis; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, multicenter, open-label, parallel-group, two-arm non-inferiority trial. Participants are assigned in a 1:1 ratio to either a PCD-CT-guided diagnostic strategy or standard invasive coronary angiography prior to TAVR evaluation.
Who Masked: Outcomes Assessor
Masking Description: An independent, blinded Clinical Events Committee will adjudicate all primary and key secondary endpoints based on medical records. The committee members will not be informed of the participants' group allocation (PCD-CT vs. ICA). The statistical analysis will also be conducted by an independent statistician blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCD-CT-Guided Diagnostic Strategy (Experimental): Participants randomized to this arm will undergo coronary artery disease (CAD) assessment using photon-counting detector computed tomography (PCD-CT). Invasive coronary angiography (ICA) will only be performed if PCD-CT shows significant CAD, defined as ≥70% diameter stenosis in vessels ≥2.5 mm or ≥50% in the left main artery.
  Interventions: Diagnostic Test: PCD-CT-Guided Diagnostic Strategy
- Standard Invasive Coronary Angiography (Active Comparator): Participants randomized to this arm will undergo routine invasive coronary angiography (ICA) as the standard of care for pre-TAVR assessment of coronary artery disease.
  Interventions: Diagnostic Test: Standard Invasive Coronary Angiography

INTERVENTIONS:
Diagnostic Test: Standard Invasive Coronary Angiography — Standard invasive coronary angiography performed routinely for all participants in this arm to assess coronary artery disease before TAVR.
  Arms: Standard Invasive Coronary Angiography
Diagnostic Test: PCD-CT-Guided Diagnostic Strategy — Participants randomized to this arm will undergo coronary artery disease (CAD) assessment using photon-counting detector computed tomography (PCD-CT). Invasive coronary angiography (ICA) will only be performed if PCD-CT shows significant CAD, defined as ≥70% diameter stenosis in vessels ≥2.5 mm or ≥50% in the left main artery.
  Arms: PCD-CT-Guided Diagnostic Strategy

SUMMARY:
The goal of this clinical trial is to determine whether a non-invasive coronary assessment strategy using photon-counting detector computed tomography (PCD-CT) is non-inferior to invasive coronary angiography (ICA) for evaluating coronary artery disease (CAD) prior to transcatheter aortic valve replacement (TAVR) in patients with severe aortic stenosis.

DETAILED DESCRIPTION:
The goal of this randomized, multicenter trial is to assess the safety and efficacy of a non-invasive diagnostic strategy using photon-counting detector computed tomography (PCD-CT) for the assessment of coronary artery disease (CAD) prior to transcatheter aortic valve replacement (TAVR), compared to the current standard of care using invasive coronary angiography (ICA).

The trial evaluates the hypothesis that a PCD-CT-guided strategy is non-inferior to routine ICA with respect to the risk of major adverse cardiovascular events (MACE) at 12 months. MACE is defined as a composite of all-cause mortality, nonfatal myocardial infarction, nonfatal stroke, urgent revascularization, or bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Severe aortic valve stenosis and indication for intervention according to current European Society of Cardiology (ESC) guidelines
* TAVR candidate
* Written informed consent

Exclusion Criteria:

* Cardiogenic shock at presentation (e.g., emergency indication for TAVR)
* Severe renal impairment with an estimated glomerular filtration rate of <30 mL/min/1.73 m²
* Life expectancy <1 year due to other severe non-cardiac disease (e.g., malignancy)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) at 12 months | 12 months after randomization
  MACE is defined as a composite of all-cause mortality, nonfatal myocardial infarction, nonfatal stroke, urgent revascularization, or bleeding events. All events will be adjudicated by an independent, blinded clinical events committee.

SECONDARY OUTCOMES:
All-cause mortality at 12 months | 12 months after randomization
  All-cause mortality is defined as death from any cause.
Cardiovascular mortality at 12 months | 12 months after randomization
  Cardiovascular death is defined as any death due to proximate cardiac or vascular cause, including death during ICA, PCD-CT, or TAVR procedures.
Nonfatal myocardial infarction at 12 months | 12 months after randomization
  Nonfatal myocardial infarction will be defined according to the Fourth Universal Definition and the VARC-3 criteria, including periprocedural and spontaneous events.
Nonfatal stroke at 12 months | 12 months after randomization
  Nonfatal stroke is defined as a neurological deficit ≥24 hours caused by ischemia or intracranial bleeding, classified per VARC-3.
Urgent revascularization at 12 months | 12 months after randomization
  Defined as unplanned hospital admission or in-hospital acute coronary syndrome requiring revascularization during the same hospitalization.
Bleeding events at 12 months | 12 months after randomization
  Bleeding events will be classified according to VARC-3 bleeding definitions, types 2 to 4.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian J Reinstadler, MD, PhD, Principal Investigator — Medical University of Innsbruck; Martin Reindl, MD, PhD, Principal Investigator — Medical University of Innsbruck
Locations (1):
- Medical University of Innsbruck, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: Undecided